CLINICAL TRIAL: NCT00720629
Title: A Phase II Study of Visilizumab for the Prevention of Graft-versus-Host Disease After Allogeneic Hematopoietic Cell Transplantation
Brief Title: Visilizumab for the Prevention of Graft-versus-Host Disease After Allogeneic Hematopoietic Cell Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MCC-15033; R01CA132197-06A2 (NIH)
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Results first posted 2014-07-04 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-04

CONDITIONS: Graft Versus Host Disease
Keywords: graft versus host disease; GVHD; allogeneic transplant; GVHD prevention; unrelated donors; mismatched unrelated donors; hematological malignancies; Leukemia; Lymphoma; Myelodysplastic Syndrome; Myelofibrosis; Aplastic Anemia; Multiple Myeloma
MeSH Terms: conditions — Graft vs Host Disease; Hematologic Neoplasms; Leukemia; Lymphoma; Myelodysplastic Syndromes; Primary Myelofibrosis; Anemia, Aplastic; Multiple Myeloma | interventions — visilizumab; Tacrolimus; Methotrexate; Antilymphocyte Serum; thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- First Study Stage: Study Treatment (Experimental): Visilizumab, Tacrolimus and Methotrexate.
  Interventions: Drug: Visilizumab; Drug: Tacrolimus; Drug: Methotrexate
- Second Study Stage: Standard Treatment (Active Comparator): Second Stage: Antithymocyte-globulin (ATG), Tacrolimus and Methotrexate. The study was closed during first stage and did not proceed to the second stage comparison to ATG in combination with tacrolimus/methotrexate as originally planned.
  Interventions: Drug: Antithymocyte globulin (ATG); Drug: Tacrolimus; Drug: Methotrexate

INTERVENTIONS:
Drug: Visilizumab — 3 mg/m^3, IV (in the vein) on day 0, prior to hematopoietic cell infusion (transplant).
  Arms: First Study Stage: Study Treatment
Drug: Tacrolimus — 0.02 mg/kg/24h (based on ideal body weight) continuous infusion (over 24 hours) beginning on day 4 after transplant up to approximately day 180 after transplant. Switch to oral tacrolimus as able. Dose adjusted based on levels. In the absence of GVHD, the dose to be tapered beginning 100 days after transplant.
  Arms: First Study Stage: Study Treatment
Drug: Methotrexate — 15 mg/m^2 intravenously (IV) on Day 1 after transplant; 10 mg/m^2 IV on Days 3, 6 and 11 after transplant.
  Arms: First Study Stage: Study Treatment
Drug: Antithymocyte globulin (ATG) — 1 mg/kg IV over 6 hours on Day 3 before transplant; 3.25 mg/kg IV over 4 hours on days 2 and 1 before transplant.
  Other Names: Thymoglobulin-ATG
  Arms: Second Study Stage: Standard Treatment
Drug: Tacrolimus — 0.03 mg/kg/24h (based on ideal body weight) continuous infusion (over 24 hours) beginning on day 3 before transplant up to approximately day 180 after transplant. Switch to oral tacrolimus as able. Dose adjusted based on levels. In the absence of GVHD, the dose to be tapered beginning 100 days after transplant.
  Arms: Second Study Stage: Standard Treatment
Drug: Methotrexate — 15 mg/m^2 IV on Day 1 after transplant; 10 mg/m^2 IV on Days 3, 6 and 11 after transplant.
  Arms: Second Study Stage: Standard Treatment

SUMMARY:
The purpose of this study was to test whether a new drug named visilizumab would decrease the severity of graft-versus-host disease in patients treated with a mismatched donor. Investigators planned to use visilizumab in combination with tacrolimus and methotrexate as the "study treatment".

DETAILED DESCRIPTION:
The protocol plan was a two stage, controlled, phase II study to assess safety and compare the grade of acute graft-versus-host disease (GVHD) with visilizumab, or Anti-thymocyte Globulin (ATG) in combination with tacrolimus + methotrexate in patients at high risk of GVHD after transplant from unrelated donors mismatched for 1-2 alleles of any type at human leukocyte antigen (HLA) A, B, C and DRB1.

The study design included two stages. The first stage of the trial was to enroll 15 patients on a single arm to be treated with "study treatment" (visilizumab, tacrolimus and methotrexate) to assess for treatment safety and exclude intolerable GVHD. The second stage of the trial was to include a random control group of patients treated with the current "standard treatment" (ATG, tacrolimus, and methotrexate) or "study treatment". The purpose of this comparison was to determine if the "study treatment" visilizumab causes less severe side effects and if it is more potent in reducing graft-versus-host disease symptoms than the "standard treatment".

ELIGIBILITY:
Inclusion Criteria:

* One of the following diagnoses with histological confirmation by the Pathology Department at H. Lee Moffitt Cancer Center:
* Acute Lymphocytic Leukemia (ALL) in complete remission 1 (CR1) with t(9:22) or t(4:11), or any ALL beyond CR1
* Acute Myelogenous Leukemia (AML) with high risk cytogenetics in CR1 as defined by Bloomfield any AML beyond CR1
* Myelodysplastic Syndrome (MDS) with International Prognostic Scoring System (IPSS) score > 1
* Chronic myelomonocytic leukemia (CMML)
* Chronic Myelogenous Leukemia (CML) with Imatinib-refractory chronic phase, or beyond chronic phase by morphology or cytogenetics
* Myelofibrosis
* Severe aplastic anemia
* Chemosensitive Non-Hodgkin's lymphoma and Hodgkin's disease that are not candidate to autologous transplant due to prior autologous transplantation
* Multiple Myeloma patient not candidate for autologous stem cell transplantation
* Karnofsky performance status ≥ 70% (adult)
* Normal organ and marrow function as defined below:
* Hepatic: Total bilirubin must be less than or equal to 2mg/dL (Gilbert and other syndromes with increased indirect bilirubin are allowed); serum transaminases must be less than two times the upper limit of normal
* Pulmonary: diffusing capacity of lung for carbon monoxide (DLCO) (corrected for Hgb), forced expiratory volume-one second (FEV1), forced vital capacity (FVC) must be greater than 50% predicted
* Cardiac: Left ventricular ejection fraction at rest must be greater than 50%
* Renal: Creatinine clearance (measured or calculated) must be equal or greater than 50 ml/min/1.73m^2

Exclusion Criteria:

* Anti thymocyte globulin (ATG) or anti T cell therapy in prior 45 days
* Splenectomized patients;
* A positive pregnancy test administered to all females of childbearing potential prior to allogeneic stem cell transplant
* Inability to comply with follow up as determined by the patient's physician
* HIV-I/II infection prior to hematopoietic stem cell (HSC) transplantation, confirmed by nucleic acid test (NAT)
* Uncontrolled bacterial or fungal infection
* History of documented invasive aspergillosis or cytomegalovirus (CMV) pneumonia
* Presence of any of the following comorbid conditions:
* History of myocardial infarction
* Congestive heart failure (even if symptomatically controlled)
* Peripheral vascular disease (including intermittent claudication or history of bypass for arterial insufficiency)
* Untreated thoracic or abdominal aneurysm (6cm or more)
* History of any cerebrovascular accident including transient ischemic attacks
* Dementia
* History of peptic ulcer disease requiring treatment
* Connective tissue/rheumatologic disorders
* Diabetes unless being managed with dietary changes only
* Hemiplegia/paraplegia
* History of solid tumor excluding skin or cervical carcinoma after curative resection

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2007-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lia Perez, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Pidala J, Perez L, Beato F, Anasetti C. Ustekinumab demonstrates activity in glucocorticoid-refractory acute GVHD. Bone Marrow Transplant. 2012 May;47(5):747-8. doi: 10.1038/bmt.2011.172. Epub 2011 Aug 29. No abstract available. PMID 21874061
- See also: H. Lee Moffitt Cancer Center & Research Institute — http://www.moffitt.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at Moffitt Cancer Center between February 2008 and April 2010.
Pre-assignment Details: The study was closed during the single-arm, first stage and did not proceed to the second stage comparison to antithymocyte globulin (ATG) in combination with tacrolimus/methotrexate as originally planned.
Groups:
- First Study Stage: Study Treatment: Visilizumab, Tacrolimus and Methotrexate. All participants.
Period: Overall Study
Arm/Group | First Study Stage: Study Treatment
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: First Stage: Study Treatment. All participants.
Groups:
- First Stage: Study Treatment: Visilizumab, Tacrolimus and Methotrexate. All participants.
Arm/Group | First Stage: Study Treatment
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: years] | 36.5 [23 to 50]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade II-IV Acute Graft-versus-Host Disease (GVHD) Score at 100 Days
Description: Cumulative Incidence of Grade II-IV Acute GVHD Score at 100 Days. Investigators had planned to assess whether the grade of acute GVHD was decreased by visilizumab in combination with tacrolimus/methotrexate compared to standard treatment with thymoglobulin/tacrolimus/methotrexate after transplantation from unrelated mismatched donors, from day of transplant up to one year. Study was closed during the first treatment stage and did not proceed to the second stage treatment comparison to ATG in combination with tacrolimus/methotrexate as originally planned.
  Overall GVHD Grade: From Filipovich AH, Weisdorf D, Pavletic S, etal: National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: I. Diagnosis and Staging Working Group Report. Biology of Blood and Marrow Transplantation 11:945-955 (2005). Grade I: Skin Stage 1-2, Liver Stage 0, Gut State 0; Grade II: Skin Stage 3 or, Liver Stage 1 or, Gut Stage 1; Grade II
Time Frame: 100 days
Population: All participants
Measure: Number; unit: participants
Arm/Group | First Study Stage: Study Treatment
Number analyzed (Participants) | 8
participants
  Grade II-IV Acute GVHD | 8
  Grade I-II Acute GVHD | 6
  Grade III-IV Acute GVHD | 2

2. Secondary Outcome: Incidence of Epstein-Barr Virus (EBV) Reactivation
Description: Number of participants who reactivated EBV. Patients had their plasma tested once weekly using the TaqMan polymerase chain reaction (PCR) for quantitative determination of EBV-DNA for 6 weeks. Plasma levels > 1000 copies per ml plasma were scored as positive.
Time Frame: 3 months
Population: All participants
Measure: Number; unit: participants
Arm/Group | First Study Stage: Study Treatment
Number analyzed (Participants) | 8
participants | 6

3. Secondary Outcome: Incidence of Rituximab Response to Reactivated EBV Without PTLD
Description: Participants who developed plasma EBV-DNA of >1000 copies/mL on any tests received rituximab.
  Incidence of Rituximab Response: Reactivated EBV participants whose plasma titers cleared after rituximab, without post-transplant lymphoproliferative disorder (PTLD).
Time Frame: 100 days
Population: Reactivated EBV participants
Measure: Number; unit: participants
Arm/Group | First Study Stage: Study Treatment
Number analyzed (Participants) | 6
participants | 6

4. Secondary Outcome: Overall Survival (OS)
Description: Median OS in days. Survival was measured from the time of transplant to the time of death.
Time Frame: At 2 years and 5 years
Population: Participants who had died by Year 2 and additional participants who had died by Year 5.
Measure: Median (Full Range); unit: days
Groups:
- 2 Year Analysis Group; 5 Year Analysis Group: First Study Stage: Study Treatment. Visilizumab, Tacrolimus and Methotrexate.
Arm/Group | 2 Year Analysis Group | 5 Year Analysis Group
Number analyzed (Participants) | 6 | 2
days | 197 [150 to 643] | 1803 [1791 to 1816]

5. Secondary Outcome: Pharmacodynamics of Visilizumab - Test 1
Description: Mean Cmax (±SD)
Time Frame: At 1 - 2 hours
Population: All participants
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | First Study Stage: Study Treatment
Number analyzed (Participants) | 8
ng/mL | 1564 (428)

6. Secondary Outcome: Pharmacodynamics of Visilizumab - Test 2
Description: Mean terminal half-life (±SD)
Time Frame: Up to 205 hours
Population: All participants
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | First Study Stage: Study Treatment
Number analyzed (Participants) | 8
hours | 157 (48)

ADVERSE EVENTS:
Time Frame: 5 years
Description: The time of administration of visilizumab on Day 1 through Day 360. Per protocol, expected transplant/GVHD-related (other than serious) adverse event details were not tabulated in the same manner as serious adverse events.
Arm/Group | First Stage: Study Treatment
Serious Adverse Events (participants affected / at risk) | 8/8
Other Adverse Events (participants affected / at risk) | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | First Stage: Study Treatment (N=8)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Hemorrhage, GI - Colon (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Febrile neutropenia (Infections and infestations) | 2
Infection - Blood (Infections and infestations) | 1
Infection - Bronchus (Infections and infestations) | 1
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other - pseudomonas pneumonia (Respiratory, thoracic and mediastinal disorders) | 1

LIMITATIONS AND CAVEATS:
Study closed early during the first stage, did not proceed to the second stage comparison as planned. Investigators exercised right to close the study prematurely for lack of efficacy, although no protocol-defined end points had been met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes